CLINICAL TRIAL: NCT06715202
Title: Effect of Educatıon Gıven To Patıents Wıth Ureteral Stent (Dj) Insertıon On Postoperatıve Symptom Management And Qualıty of Lıfe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muazzez Merve TORAMAN, Research Assistant, Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Muazzez Merve TORAMAN
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Ureteral Calculi
Keywords: Ureteral Stent (DJ), Symptom Management, Quality of Life
MeSH Terms: conditions — Ureteral Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Patient Education Booklet (Experimental): Patients will be informed about URS, DJ stents and possible problems in the early postoperative period with an education booklet and the patient's questions will be answered.
  Interventions: Procedure: Patient Education Booklet

INTERVENTIONS:
Procedure: Patient Education Booklet — Before the surgery, a personal information form and the SF-36 Quality of Life Scale will be filled out. The educational content regarding the problems that these patients may encounter with the DJ stent after the surgery until they are discharged will be explained in sections and the patients' questions will be answered. When the patient comes to the hospital for DJ stent removal 4 weeks after discharge, the Ureteral Stent Symptom 1st Questionnaire and the SF-36 Quality of Life Scale will be filled out while the DJ stent is in place. The Ureteral Stent Symptom 2nd Questionnaire and the SF-36 Quality of Life Scale will be applied 4 weeks after the stent is removed. The education booklet will be prepared by the researchers in accordance with the recommendations of the European Association of Urology and the relevant literature.

SUMMARY:
The data of the randomized controlled experimental study were collected at the Urology Clinics of Atatürk University Health Practice and Research Hospital between April and November 2022. The study sample consisted of 162 patients (82 in the training group, 80 in the control group) who were selected by simple random sampling method and met the inclusion criteria for the study.

DETAILED DESCRIPTION:
Ureteral stents have been widely used in many urological procedures since their use was published by Zimskind in 1967 and Finley's use of the modern double J (DJ) stent in 1978. Ureterorenoscopy (URS) is a popular method used frequently in the diagnosis and treatment of ureteral diseases today. Apart from being performed for diagnostic purposes, URS is most commonly used to treat ureteral stones. The vast majority of ureteral stones are treated endoscopically. A Double-J (DJ) stent is often placed after ureterorenoscopy. The purpose of the stent is to prevent obstruction, renal colic, and deterioration of renal function. The fact that the DJ stent will remain in the patient for a certain period of time (approximately 3-4 weeks) causes anxiety in the patient. However, urinary system symptoms that impair the quality of life are observed in approximately 80% of patients who have a DJ stent. These symptoms include frequent urination (50-60%), urgency (57-60%), pain during urination (40%), incomplete voiding (76%), flank pain (19-32%), suprapubic pain (30%), incontinence and hematuria (25%). In addition, 32% of patients with DJ stents develop sexual dysfunction. 2,3,4 Patients who have DJ stents inserted after ureteroscopy surgery need more information, support, explanation and help to cope with the effects of these symptoms in the clinic and at home. 5 In this context, it is important to provide individualized and comprehensive education that includes the home care process before and after URS. It has been determined in the literature that education given before surgical intervention reduces anxiety, pain level, complication rate and depression rate in the postoperative period and increases patient satisfaction. 6,7,8 However, it is reported that individuals should be discharged with sufficient theory and practice to meet their post-discharge care needs. Although all healthcare personnel are responsible for the discharge education of individuals and their relatives, the most important responsibility belongs to nurses.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Volunteering to participate in the study
* Having URS surgery for the first time due to stones and temporary DJ stent placement

Exclusion Criteria:

* Having URS surgery for reasons other than stones
* Having a permanent stent
* Having major hearing and vision impairment
* Using antidepressants or anxiolytics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | The universe of the study, between April and November 2022.
  Ureteral Stent Symptom Questionnaire: In 2003, Joshi and colleagues developed a special questionnaire for the assessment of quality of life and stent-related symptoms. The Ureteral Stent Symptoms Questionnaire (USSQ), a validated tool that assesses symptoms and quality of life, was validated in Turkish by Yılören and colleagues in 2017. The USSQ was originally designed as a 38-item questionnaire with 33 Likert-type questions and 5 more descriptive items organized into six main areas. This questionnaire provides a comprehensive assessment of urinary symptoms, general health, pain, sexual health, work performance, and other additional problems related to ureteral stents

CONTACTS AND LOCATIONS:
Locations (1):
- Muazzez Merve TORAMAN, Erzurum, Turkey (Türkiye)